CLINICAL TRIAL: NCT02376010
Title: Rivaroxaban Versus Warfarin in the Evaluation of Progression of Coronary Calcium
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Responsible Party: Principal Investigator, Matthew J. Budoff, Principal Investigator, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21429
Record Dates: First submitted 2015-02-24; First posted 2015-03-03 (Estimated); Results first posted 2021-07-22 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Atherosclerosis
Keywords: atherosclerosis; coronary artery disease; cardiac CT; computed tomographic angiography
MeSH Terms: conditions — Atherosclerosis; Coronary Artery Disease | interventions — Rivaroxaban; Warfarin

STUDY DESIGN:
Intervention Model Description: randomized controlled trial, with blinded randomization to one of two groups.
Oversight: Data Monitoring Committee: No

ARMS (2):
- rivaroxaban (Active Comparator): rivaroxaban will be given to this cohort, once daily orally (15 or 20 mg, depending on GFR)
  Interventions: Drug: rivaroxaban
- warfarin (Active Comparator): warfarin orally once a day, titrated to INR of 2-3
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: rivaroxaban
  Arms: rivaroxaban
Drug: Warfarin
  Arms: warfarin

SUMMARY:
Current oral anti-coagulation for atrial fibrillation is most commonly performed with warfarin. Warfarin is a vitamin K antagonist that has been shown in non-randomized trials to increase vascular calcification. Increased vascular calcification has been tied to increased cardiovascular events (CVE). This study will randomize patients currently taking warfarin to either continue on warfarin or be switched to rivaroxaban. Rivaroxaban is an oral anti-coagulant that works by inhibiting Factor Xa, and has no interaction with vitamin K. This study is a randomized, open label study that will randomize 120 patients and have them undergo blood tests and a calcium scan at baseline, and again after 12 months. Patients will be seen quarterly for examinations, safety checks and supply of rivaroxaban, as well as follow up INR testing for warfarin.

DETAILED DESCRIPTION:
Rivaroxaban is a novel oral direct factor Xa inhibitor that has been shown to reduce the risk of stroke in a similar population in comparison with warfarin. The rate of myocardial infarction was 9% lower in the rivaroxaban group than in the warfarin group in the Rocket AF study and similarly the myocardial infarction rate was 12% lower in the apixaban group in Aristotle, but the difference was not significant in either trial. The potential of long term benefit by avoiding VKA therapy may be much greater for a CV event reduction. The study proposed will evaluate markers of CAC progression and atherosclerosis development, which have long term outcome data supporting that slowing these processes will be associated with lower CV events.

ELIGIBILITY:
Key Inclusion Criteria:

1. Eligible patients with atrial fibrillation at enrollment or two or more episodes of atrial fibrillation or flutter, as documented by electrocardiography, at least 2 weeks apart in the 12 months before enrollment
2. Age 18-84
3. On Warfarin for 6 months prior to enrollment at a stable dose.
4. Willingness to participate in the study and ability to sign informed consent
5. Minimum CAC score of 10

Key Exclusion Criteria:

1. Atrial fibrillation due to a reversible cause, moderate or severe mitral stenosis, or conditions other than atrial fibrillation that require anticoagulation (e.g., a prosthetic heart valve)
2. Prior apixaban, dabigatran, rivaroxaban use.
3. A need for aspirin at a dose of >165 mg a day or for both aspirin and clopidogrel,
4. Renal insufficiency (serum creatinine level of 12.5 mg per deciliter or calculated creatinine clearance of <50 ml per minute).
5. Serious bleeding event in the previous 6 months or a high risk of bleeding (eg, active peptic ulcer disease, a platelet count of <100,000/mm3 or hemoglobin level of <10 g/dL, stroke within the previous 10 days, documented hemorrhagic tendencies, or blood dyscrasias)
6. Weight in excess of 325 pounds
7. Resting hypotension (systolic blood pressure of <90mmHg) or resting hypertension (systolic blood pressure of >170mmHg or diastolic blood pressure of >110 mmHg).
8. History of active malignancy requiring concurrent chemotherapy.
9. Any unstable medical, psychiatric, or substance abuse disorder that in the opinion of the principal investigator is likely to affect the subject's ability to complete the study.
10. Known allergy to iodinated contrast material
11. Pregnancy or breast feeding

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2015-04-02 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Los Angeles Biomedical Research Institute, Torrance, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Rivaroxaban: rivaroxaban will be given to this cohort, once daily orally (15 or 20 mg, depending on GFR)
  rivaroxaban
- Warfarin: warfarin orally once a day, titrated to INR of 2-3
  Warfarin
Period: Overall Study
Arm/Group | Rivaroxaban | Warfarin
Started | 55 | 55
Completed | 46 | 51
Not Completed | 9 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rivaroxaban | Warfarin | Total
Number analyzed (Participants) | 55 | 55 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 41 | 83
  >=65 years | 13 | 14 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (10) | 60 (11) | 61 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 33
  Male | 39 | 38 | 77
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 11 | 22
  White | 43 | 42 | 85
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 55 | 55 | 110

OUTCOME MEASURES:

1. Primary Outcome: Coronary Artery Calcium (Serial Calcium Scans)
Description: serial calcium scans
Time Frame: 1 year
Population: patients completed second scan with interpretable data
Measure: Median (Inter-Quartile Range); unit: mm cubed
Arm/Group | Rivaroxaban | Warfarin
Number analyzed (Participants) | 46 | 51
mm cubed | 26.3 [4.5 to 61.5] | 40.5 [9.6 to 97.3]

2. Secondary Outcome: Atherosclerotic Plaque (Measures of Total Atherosclerosis Plaque on Serial CCTA)
Description: measures of total atherosclerosis plaque on serial CCTA
Time Frame: 1 year
Population: volume of plaque in patients completing study
Measure: Median (Inter-Quartile Range); unit: mm cubed
Arm/Group | Rivaroxaban | Warfarin
Number analyzed (Participants) | 46 | 51
mm cubed | 20.1 [0 to 45] | 30.1 [2 to 72]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Rivaroxaban | Warfarin
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/51
Other Adverse Events (participants affected / at risk) | 1/46 | 2/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rivaroxaban (N=46) | Warfarin (N=51)
minor bleeding (Blood and lymphatic system disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-02): https://cdn.clinicaltrials.gov/large-docs/10/NCT02376010/Prot_SAP_000.pdf